CLINICAL TRIAL: NCT04713410
Title: Comparison of Relapse Rate After 12 Weeks Verses 20 Weeks Steroid Therapy for the Management of First Episode of Steroid Sensitive Nephrotic Syndrome: A Randomized Control Trial at Children Hospital, Pakistan Institute of Medical Sciences, Islamabad
Brief Title: Comparison of Relapse Rate After 12 Weeks Verses 20 Weeks Steroid Therapy for the Management of First Episode of Steroid Sensitive Nephrotic Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shaheed Zulfiqar Ali Bhutto Medical University (Other)
Responsible Party: Principal Investigator, Dr Nighat Haider, Assistant Professor, Shaheed Zulfiqar Ali Bhutto Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: No.F.1-1/2015/ERB/SZABMU/465
Record Dates: First submitted 2021-01-14; First posted 2021-01-19 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Steroid-Sensitive Nephrotic Syndrome
Keywords: Nephrotic Syndrome, steroid response, relapse
MeSH Terms: conditions — Nephrotic Syndrome; Recurrence | interventions — Prednisolone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Steroids will be given for short duration of time i-e 12 weeks
  Interventions: Drug: Prednisolone
- Group B (Active Comparator): Steroid will be given for longer duration i-e 20 weeks
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Prednisolone — Regimen will be to administer prednisolone as a single dose of 60 mg/m2 once daily for 6 weeks, then 40 mg/m2 on alternate day.

SUMMARY:
All children from 1 to 8 years of age, diagnose with nephrotic syndrome for the first time will be divided into two groups. One group will be given steroids for 12 weeks and other group will receive steroid for 20 weeks. During the 1 years after completion of steroid course patients will be monitor for the episodes of relapse in both group.

DETAILED DESCRIPTION:
All children from 1 to 8 years of age, diagnose with nephrotic syndrome for the first time, at Pakistan Institute of Medical Sciences, Islamabad, from December 2020 to December 2022 will be included in the study.

Sample size was calculated by using WHO sample size calculator keeping level of significance 5%, power of test 90%, P1 21.6%7 and P2 59.3%8. The sample size is turned out to be 34 patients in each group with total of 68 patients.

The patients fulfilling the inclusion criteria will be registered at our nephrology clinic. Patients' bio data along with history and examination will be recorded on a proforma. They will be divided in two groups designated as A and B. Group A will receive steroid for 12 weeks and group B for 20 weeks. For group A regimen will be to administer prednisolone as a single dose of 60 mg/m2 once daily for 6 weeks, then 40 mg/m2 on alternate day for another 6 weeks and then stop. For group B prednisolone will be given as a single dose of 60 mg/m2 once daily for 6 weeks, then 40 mg/m2 on alternate day for another 6 weeks with tapering of 25% of alternate day dose fortnightly. Outcome will be measured in terms of number of relapses in the subsequent 1 years after stopping steroids.

For treatment of relapse Prednisolone will be given in the dose of 60 mg/m2 once daily till urine protein is negative or trace for 3 consecutive days, then 40 mg/m2 on alternate day for 1 month then stop. In case of frequent relapses and steroid dependent cases, relapses will be treated as follows; prednisolone 60 mg/m2 on alternate day till urine protein will be negative for 5days then 40 mg/m2 on alternate day for 1 month then with tapering at the rate of 5 mg fortnightly.

Children with congenital and infantile nephrotic syndrome, persistent hypertension, gross haematuria, family history of nephrotic syndrome and age below 1 year and above 8 years will be excluded from study.

After approval of study from ethical review board, informed consent will be taken from parents. The data obtained will be analyzed using SPSS version 20. The t test will be applied for comparison of mean and chi sqare test for comparison of percentages. The p value less than .05 will be taken as significant.

ELIGIBILITY:
Inclusion Criteria:

* Children 1 to 8 years of age,
* Diagnose with nephrotic syndrome for the first time
* Steroid sensitive nephrotic syndrome

Exclusion Criteria:

* Steroid resistant nephrotic syndrome
* Steroid dependent nephrotic syndrome
* Syndromic Children
* Children with other co morbidities

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Estimated)
Dates: Start 2020-12-22 (Actual); Primary Completion 2022-09-04 (Estimated); Study Completion 2023-09-04 (Estimated)

PRIMARY OUTCOMES:
Relapse rate | 2 years
  Relapse rete

CONTACTS AND LOCATIONS:
Locations (1):
- Pakistan Institute of Medical Sciences, Islamabad, Capital, Pakistan